CLINICAL TRIAL: NCT03759015
Title: Evaluation of Health Education Theater
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1341383
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Community Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health education (Other): This arm's subjects are tasked to create an original 10-minute theater that is required to use the guidelines about physical activity and diet/nutrition.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — All subjects are tasked to create an original 10-minute theater about physical activity and diet/nutrition.

SUMMARY:
This study evaluates the feasibility and the potential positive health impacts of a novel "health education theater," which will task participants of a health education program to create an original 10-minute theater that is required to use the health guidelines about physical activity and diet/nutrition. The outcomes include the changes in (a) knowledge about these guidelines, (b) compliance to these guidelines, (c) health related quality of life, and (d) self-perception well-being measures such as self-esteem and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* University of California (UC) Davis students who register for the course entitled " Health Education Theater," to be held during the 2019 Spring Quarter, i.e., from April 2019 to June 2019.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Individuals who are not compliant to this project's guideline of health limitations. Under this project guideline, absences due to health limitations are not expected to exceed 3 days maximum in addition to standard class policy during the quarter. As long as a subject is compliant to this project guideline and the additional accommodations authorized by the UC Davis Student Disability Center (SDC), any student (including a pregnant woman student and a student with a disability) can participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge about the health guidelines regarding physical activity | baseline, immediately post-intervention, 6 months post-intervention, 12-months post-intervention
  Knowledge about the guidelines regarding physical activity assessed via survey questionnaire. This outcome is dichotomous, either 0 or 1, representing a survey respondent's knowledge about the guideline is incorrect or correct, respectively. This guideline is set by the UC Davis Health Education and Promotion (HEP) (https://shcs.ucdavis.edu/wellness/physical-activity).
Change in knowledge about the health guidelines regarding diet/nutrition | baseline, immediately post-intervention, 6 months post-intervention, 12-months post-intervention
  Knowledge about the guidelines regarding diet/nutrition assessed via survey questionnaire. This outcome is dichotomous, either 0 or 1, representing a survey respondent's knowledge about the guideline is incorrect or correct, respectively. This guideline is set by the UC Davis Health Education and Promotion (HEP) (https://shcs.ucdavis.edu/fruits-andveggies).
Change in compliance about the health guidelines regarding physical activity | baseline, immediately post-intervention, 6 months post-intervention, 12-months post-intervention
  Compliance about the guidelines regarding physical activity assessed via survey questionnaire. This outcome is dichotomous, either 0 or 1, representing a survey respondent is non-compliant or compliant to the guideline, respectively. This guideline is set by the UC Davis Health Education and Promotion (HEP) (https://shcs.ucdavis.edu/wellness/physical-activity).
Change in compliance about the health guidelines regarding diet/nutrition | baseline, immediately post-intervention, 6 months post-intervention, 12-months post-intervention
  Compliance about the guidelines regarding diet/nutrition assessed via survey questionnaire. This outcome is dichotomous, either 0 or 1, representing a survey respondent is non-compliant or compliant to the guideline, respectively. This guideline is set by the UC Davis Health Education and Promotion (HEP) (https://shcs.ucdavis.edu/fruits-andveggies).
Change in health related quality of life | baseline, immediately post-intervention, 6 months postintervention, 12-months post-intervention
  Health related quality of life will be measured with the unit of utility (ranging from 0 to 100), which will be derived with the established method of visual analogue scale following EuroQol Group (Health Policy. 1990;16(3):199-208).
Change in self-esteem | baseline, immediately post-intervention, 6 months postintervention, 12-months post-intervention
  Self-esteem will be measured by the established method of "the Rosenberg's self-esteem scale," ranging from 10 to 40 (Rosenberg M. Society and the Adolescent Self-Image. Princeton, NJ, Princeton University Press, 1965).
Change in self-efficacy | baseline, immediately post-intervention, 6 months postintervention, 12-months post-intervention
  Self-efficacy will be measured by the established method of "the Generalized self-efficacy scale," ranging from 10 to 40 (Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, &M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, England: NFER-NELSON.).

SECONDARY OUTCOMES:
Economic efficiency of the intervention | 60 years after the end of the intervention based on a simulation analysis
  Return on investment (ROI) of the intervention based on a simulation analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/an-evaluation-of-the-health-education-theater-course-151816/